CLINICAL TRIAL: NCT04402606
Title: DERMACLIC : Study on Skin Toxicities Induced by Cancer Treatments
Brief Title: Study on Skin Toxicities Induced by Cancer Treatments
Acronym: DERMACLIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A0872-55
Record Dates: First submitted 2020-04-29; First posted 2020-05-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor, Adult; Breast Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation on skin toxicities (Experimental): This evaluation consists on a clinical examination of the skin and the realization of the cutaneous measurements of reference on 4 sites frequently exposed to the cutaneous toxicities: face, neckline, palms of the hands and soles of the feet.
  Interventions: Other: Evaluation on skin toxicities

INTERVENTIONS:
Other: Evaluation on skin toxicities — Measurements will be carried out using specific tools, such as the cutaneous ultrasound system (measurement of the skin layers thicknesses, the cutometer (measurement of the elasticity of the skin), the corneometer (measurement of the hydration of the skin), the pH meter (measuring the pH of the skin), the colorimeter (measuring the color of the skin), the tewameter (measuring the insensible loss of water), the sebometer (measuring sebum).

SUMMARY:
The skin toxicities will be evaluated on patient (male or female) with an indication of cancer treatment in the case of solid tumor of the breast, or lung.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, male or female, aged 18 years and older, with a solid tumor breast or lung, localized, locally advanced or not, metastatic or not;
2. Patient in medical oncology consultation requiring systemic anti-tumor therapy (chemotherapy, targeted therapy, hormone therapy, immunotherapy) in neo-adjuvant, adjuvant or metastatic;
3. Treatment planned for a minimum period of 3 months (from the date of inclusion);
4. Having a social security protection;
5. Signed informed consent form of the study.

Exclusion Criteria:

1. Patient treated for lymphoma, leukemia or inflammatory breast cancer ;
2. Patient with a solid tumour which location is other than breast or lung;
3. Patient with a tumor wound ;
4. Patient with a general condition > 2 at baseline (ECOG classification) ;
5. Patient receiving anti-tumor treatment with radiotherapy exclusively or associated with concomitant radiotherapy ;
6. Patient unable to receive information about the study and to give consent ;
7. Persons deprived of liberty or guardianship ;
8. Impossible submission to study procedures for geographical or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Estimate the rates of severe skin toxicities (grade 2) induced by cancer treatments, at 8 months after the start of treatment. | 8 months
  Severity of cutaneous toxicities at 8 months after the start of treatment (grade > 2 according to the NCI-CTCAE classification version 4.03), induced by the anticancer treatments.

SECONDARY OUTCOMES:
Evaluate the thickness, firmness, tone, viscosity of the skin in case of skin toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. A cutaneous ultrasound system will be used to evaluate thickness of the skin and a cutometer will be used to evaluate firmness, tone and viscosity of the skin. The measurement in millimeters will be used to assess this outcome measure.
Evaluate skin color in case of skin toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. A colorimeter will be used to evaluate skin color. No unit will be used to assess this outcome measure.
Evaluate the skin pH in case of skin toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. A pHmeter will be used to evaluate skin pH. No unit will be used to assess this outcome measure
Evaluate the temperature in case of skin toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. Thermometer will be used to evaluate temperature of the skin. The measurement in degrees Celsius will be used to assess this outcome measure.
Evaluate the quantity of sebum in case of toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. Sebumeter will be used to evaluate quantity of sebum of the skin. The measurement in microgram/centimeter^2 will be used to assess this outcome measure
Evaluate plantar supports in case of toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. Podobarometric platform will be used to evaluate plantar supports. The measurement in N/Centimeter^2 will be used to assess this outcome measure.
Evaluate Skin hydration rate in case of skin toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. Corneometer will be used to evaluate skin hydration rate. No unit will be used to assess this outcome measure.
Evaluate skin elasticity index in case of toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. Cutometer will be used to evaluate skin elasticy. No unit will be used to assess this outcome measure.
Evaluate insensitive loss of water in case of toxicities | 8 months
  The assessments will be performed at day 0 (before the start of the study) and at 1 month (M1), M2, M3, M4 and M8 after the start of treatment. Tewameter will be used to evaluate insensitive loss of water. The measurement in gram/meter^2/hour will be used to assess this outcome measure.
Evaluate variation rate of thickness, firmness, tone, viscosity of the skin over the course of the study | 8 months
  A cutaneous ultrasound system will be used to evaluate thickness of the skin and a cutometer will be used to evaluate firmness, tone and viscosity of the skin. The measurement in millimeters will be used to assess this outcome measure. Variations of thickness, firmness, tone, viscosity of the skin will be calculated according to results obtained at M1, M2,M3, M4 and M8. Results will be compared to initial measures at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of skin color over the course of the study | 8 months
  A colorimeter will be used to evaluate skin color. No unit will be used to assess this outcome measure. Variations of skin color will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of skin pH over the course of the study | 8 months
  A pHmeter will be used to evaluate skin pH. No unit will be used to assess this outcome measure. Variations of pH of the skin will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage
Evaluate variation rate of skin temperature over the course of the study | 8 months
  A thermometer will be used to evaluate skin temperature. The measurement in degrees Celsius will be used to assess this outcome measure. Variations of temperature of the skin will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of skin sebum quantity over the course of the study | 8 months
  A sebumeter will be used to evaluate quantity of sebum of the skin. The measurement in microgram/centimeter^2 will be used to assess this outcome measure. Variations of quantity of sebum of the skin will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of plantar supports over the course of the study | 8 months
  A podobarometric platform will be used to evaluate plantar supports. The measurement in N/Centimeter^2 will be used to assess this outcome measure. Variations of plantar supports will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of skin hydration over the course of the study | 8 months
  A corneometer will be used to evaluate skin hydration rate. No unit will be used to assess this outcome measure. Variations of skin hydration of the skin will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of skin elasticity over the course of the study | 8 months
  A cutometer will be used to evaluate skin elasticy. No unit will be used to assess this outcome measure. Variations of elasticity of the skin will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate variation rate of insensitive loss of water of the skin over the course of the study | 8 months
  A tewameter will be used to evaluate insensitive loss of water. The measurement in gram/meter^2/hour will be used to assess this outcome measure. Variations of insensitive loss of water of the skin will be calculated according to results obtained at M1, M2,M3,M4 and M8. Results will be compared to initial measure at day 0. Variation rate will be estimated in percentage.
Evaluate the consequences of cutaneous toxicities on the patient's therapeutic scheme (hold, dosage reduction, change of molecule); | 8 months
  Number of treatment interruptions or dose changes related to skin toxicities;
To evaluate the quality of life of patients at 8 months; | 8 months
  A questionnaire (Medical Outcome Study Short Form - 36 (MOS SF-36) will be completed by patients. This is a scale allowing to assess health regardless of causal pathology, gender, age and treatment, which is related to patients level of well-being. A score from 0 (poor quality of life) to 100 (very good quality of life) will be given;
Define patient profiles likely to develop severe cutaneous toxicity during their anticancer treatment; | 8 months
  During these assessments, a census of skin toxicities (grade >2) will be carried out according to the NCI-CTCAE version 4.03 classification, and the patient's medical record will be analyzed to determine the predictors of skin toxicities.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie, Paris, France